CLINICAL TRIAL: NCT00636623
Title: Comparison of Pilates Exercises and Connective Tissue Massage in Females With Fibromyalgia
Brief Title: Comparison of Exercise and Massage in Fibromyalgia
Acronym: FM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Gamze Ekici, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ekici - 2; ISRCTN12345678
Record Dates: First submitted 2008-03-07; First posted 2008-03-14 (Estimated); Last update posted 2008-03-14 (Estimated); Status verified 2008-03

CONDITIONS: Fibromyalgia
Keywords: Pilates Exercises; Connective Tissue Massage
MeSH Terms: conditions — Fibromyalgia | interventions — Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Other): Pilates exercises
  Interventions: Other: Pilates exercises
- 1 (Other): Connective tissue massage
  Interventions: Other: Connective tissue massage

INTERVENTIONS:
Other: Pilates exercises — 15 FM patients participated in the PE programme three times a week during a 4-week period
  Other Names: No drug name
  Arms: 2
Other: Connective tissue massage — 21 patients received CTM, three times a week during a 4-week period
  Arms: 1

SUMMARY:
The present study was designed to analyse and compare the effects of Pilates exercises and connective tissue massage in terms of pain intensity, pain pressure threshold and tolerance, anxiety, progress, and health related quality of life in females with fibromyalgia (FM)

DETAILED DESCRIPTION:
Treatment of FM is difficult. Conventional treatments do not appear to be managing the problem effectively and this has led to other forms of treatment. The aim of treating FM is to decrease pain and increase function by means of a multimodal therapeutic strategy, which, in most cases, includes pharmacological and non-pharmacological interventions. In the literature on non-pharmacological treatment approaches for FM, different managements are described, such as exercise, electrotherapy, patient education, self-management programmes, massage techniques, cryotherapy, and acupuncture. There are a number of reasons why patients choose these complementary and alternative medicine approaches, including dissatisfaction with conventional treatments or concerns over the toxicity of drugs. However, there is no consensus about which treatment approach is the best.The current randomised controlled trial was undertaken as a first pilot study to assess and compare the effectiveness of Pilates exercises, an active-group therapy, and connective tissue massage, a passive-personalised therapy, in the management of FM in females.

ELIGIBILITY:
Inclusion Criteria:

* being female
* being over 25 years old
* meeting the criteria for FM as defined by the American College of Rheumatology
* having pain in the neck and shoulder region
* never having been treated for FM.

Exclusion Criteria:

* infection
* fever or an increased tendency to bleed
* severe physical impairment
* inflammatory diseases
* cardiopulmonary disorders
* uncontrolled endocrine disorders
* allergic disorders
* pregnancy
* malignancy
* severe psychiatric illnesses
* factors known to affect autonomic function
* medication usage

Ages: 25 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2006-11; Primary Completion 2007-07 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale, algometry, State-Trait Anxiety Inventory (STAI), Fibromyalgia Impact Questionnaire, and Nottingham Health Profile were used at baseline and at the end of the treatments. | For All measurements aproximately 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Gamze Ekici, PhD, Principal Investigator — Pamukkale University; Turkan Akbayrak, Assoc. Prof., Study Director — Hacettepe University; Edibe Yakut, Prof, Study Director — Hacettepe University; Naciye Vardar, MsC, Study Director — Hacettepe University; Yavuz Yakut, Prof, Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)